CLINICAL TRIAL: NCT02262546
Title: A Double-blind, Randomised, Placebo Controlled Study With Two Sequential Two-way Cross-over Parts to Demonstrate That the Influence of Pramipexole up to 4.5 mg Daily on the QT Interval of the ECG in Healthy Male and Female Volunteers is Comparable With Placebo, With a Positive Control (Two-way Cross-over Moxifloxacin Versus Placebo)
Brief Title: Influence of Pramipexole on the QT Interval of the ECG in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 248.545
Record Dates: First submitted 2014-10-09; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Tablets; Moxifloxacin

ARMS (4):
- Pramipexole (Experimental)
  Interventions: Drug: Pramipexole extended-release (ER) tablets; Drug: Pramipexole immediate-release (IR) tablets
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin
- Pramipexole Placebo (Placebo Comparator)
  Interventions: Drug: Pramipexole Placebo
- Moxifloxacin Placebo (Placebo Comparator)
  Interventions: Drug: Moxifloxacin Placebo

INTERVENTIONS:
Drug: Pramipexole extended-release (ER) tablets
  Arms: Pramipexole
Drug: Pramipexole immediate-release (IR) tablets
  Arms: Pramipexole
Drug: Moxifloxacin
  Arms: Moxifloxacin
Drug: Pramipexole Placebo
  Arms: Pramipexole Placebo
Drug: Moxifloxacin Placebo
  Arms: Moxifloxacin Placebo

SUMMARY:
The objective of the study is to assess that pramipexole does not prolong the QT interval more than placebo

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study need to be healthy males or females 21 to 50 years of age
* Body mass index (BMI) ranging from 18.5 to 29.9 kg/m2
* Signed written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (≤ 30 days prior to administration or during the trial)
* Heavy smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≥ 100 mL within four weeks prior to administration or during the trial)
* Any deviation of a laboratory value that is considered to be of clinical relevance
* Excessive physical activities within the last week before the trial or during the trial
* Hypersensitivity to pramipexole, moxifloxacin and/or related drugs of these classes
* Supine blood pressure at screening of systolic < 100 mmHg and diastolic < 60 mmHg
* Heart rate at screening of > 80 beats per minute (bpm) or < 40 bpm
* Any screening ECG value outside of the reference range of clinical relevance including, but not limited to Pulse Rate interval > 220 ms, QRS interval > 115 ms, QTcB or QTcF > 450 ms, or QT (uncorrected) > 470 ms
* Subjects involved in passenger transport or operation of dangerous machines

For Female Subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (adequate contraception: e.g. sterilization, intrauterine device, oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-05; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Mean of the individually heart rate corrected QT interval (QTcI) values | 1 to 4 hours after dosing on day 21

SECONDARY OUTCOMES:
Mean of the QTcI values | 1 to 4 hours after dosing at day 12
QTcI at any point in time | between 1 and 7 hours after dosing at day 12 and day 21